CLINICAL TRIAL: NCT06514040
Title: Nebulized Dexmedetomidine Versus Oral Sumatriptan for Treatment of Post-Dural Puncture Headache Following Caesarian Section (Randomized Comparative Study)
Brief Title: Nebulized Dexmedetomidine Versus Oral Sumatriptan in Treatment of Post Dural Puncture Headache in Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fayoum University Hospital (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Hamed, Assistant professor, Fayoum University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M684
Record Dates: First submitted 2024-05-09; First posted 2024-07-23 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Post-Dural Puncture Headache
MeSH Terms: conditions — Post-Dural Puncture Headache | interventions — Dexmedetomidine; Sumatriptan

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Precedex group (Active Comparator): 1- Inhaled Dexmedetomidine group (Group D, n= 24): will receive nebulization of 1 µg/kg dexmedetomidine (Precedex, Dexmedetomidine HCl 100 µg/mL, Pfizer Inc.) diluted in 4 mL 0.9% saline twice daily starting from the PDPH diagnosis time. The intervention will be continued until achieving a VAS score ≤ 3 and Lybecker classification score < 2 or for a maximum of 48 hours when occurrence of side effects in form of hypotension, bradycardia, nausea stop the medication and give supportive treatment.
  Interventions: Drug: Precedex
- Sumatriptan group (Active Comparator): 2- Oral sumatriptan group (Group S, n= 24): sumatriptan 25 mg every 8 hours orally when occurrence of side effects in form of paresthesia, dizziness and chest tightness stop the medication.
  Interventions: Drug: Sumatriptan 25 mg

INTERVENTIONS:
Drug: Precedex — Dexmedetomidine (Precedex) is a highly selective alpha 2 adrenoreceptor agonist which produce sedation, anxiolysis, analgesia, and decreasing inflammatory response to anaesthesia and surgical procedure.
  Arms: Precedex group
Drug: Sumatriptan 25 mg — Sumatriptan (Imigran) is a selective serotonin receptor agonist. It works by narrowing blood vessels in the brain, stopping pain signals from being sent to the brain, and blocking the release of certain natural substances that cause pain (as substance -p), nausea, and other symptoms of migraine
  Arms: Sumatriptan group

SUMMARY:
comparison between oral sumatriptan and Nebulized Dexmedetomidine in Post Dural Puncture Headache in Cesarean Section

DETAILED DESCRIPTION:
A total of 48 patients will be randomly chosen to receive either inhaled dexmedetomidine (Group D, n= 24) or oral sumatriptan (Group S, n= 24) by a random sequence number generated by the computer kept in sealed envelopes. Those envelopes will be opened once the patient is recruited and participants will receive either inhaled dexmedetomidine or oral sumatriptan as per the envelope. Data collectors will be blinded to the type of used medication (Dexmedetomidine or Sumatriptan).

ELIGIBILITY:
Inclusion criteria:

1. Pregnant female aged between 18 and 40 years old.
2. ASA II and III undergoing elective caesarean section.
3. Diagnosed with Postdural puncture headache with visual analogue score (VAS) ≥ 4 and Lybecker classification score ≥ 2.

Exclusion criteria:

1. Patient refusal.
2. History of primary headaches such as migraine, cluster and tension headaches.
3. Hypersensitivity of dexmedetomidine or sumatriptan.
4. Hypertensive disorders of the pregnancy.
5. Contraindication to spinal anesthesia as coagulopathy or infection at site of injection.
6. Symptoms of ischemic heart disease (IHD) e.g. angina.
7. Cerebrovascular disease e.g. stroke or transient ischemic attacks (TIAs).
8. Using of Monoamine oxidase inhibitors (MAOIs) in the last 24h.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant female
Enrollment: 48 (Actual)
Dates: Start 2023-11-27 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
visual analogue scale | First 48 hours
  VAS Score from 0 to 10 where score 0 is no headache and 10 is the worst one

SECONDARY OUTCOMES:
visual analogue scale | 6 hours.
  VAS Score from 0 to 10 where score 0 is no headache and 10 is the worst one
visual analogue scale | 12 hours.
  VAS Score from 0 to 10 where score 0 is no headache and 10 is the worst one
visual analogue scale | 18 hours.
  VAS Score from 0 to 10 where score 0 is no headache and 10 is the worst one
visual analogue scale | 24 hours.
  VAS Score from 0 to 10 where score 0 is no headache and 10 is the worst one
visual analogue scale | 30 hours.
  VAS Score from 0 to 10 where score 0 is no headache and 10 is the worst one
visual analogue scale | 36 hours.
  VAS Score from 0 to 10 where score 0 is no headache and 10 is the worst one
visual analogue scale | 42 hours.
  VAS Score from 0 to 10 where score 0 is no headache and 10 is the worst one
Lybecker score | 6 hours
  Mild
  Mild:Daily activities slightly restricted. Patient is not bedridden
  No associated symptoms
  Moderate:Daily activities significantly restricted and most of the day patient is bedridden with or without associated symptoms
  Severe:Daily activities completely restricted, patient is bedridden all the day and always with associated symptoms
Lybecker score | 12 hours
  Mild
  Mild:Daily activities slightly restricted. Patient is not bedridden
  No associated symptoms
  Moderate:Daily activities significantly restricted and most of the day patient is bedridden with or without associated symptoms
  Severe:Daily activities completely restricted, patient is bedridden all the day and always with associated symptoms
Lybecker score | 18 hours
  Mild
  Mild:Daily activities slightly restricted. Patient is not bedridden
  No associated symptoms
  Moderate:Daily activities significantly restricted and most of the day patient is bedridden with or without associated symptoms
  Severe:Daily activities completely restricted, patient is bedridden all the day and always with associated symptoms
Lybecker score | 24 hours
  Mild
  Mild:Daily activities slightly restricted. Patient is not bedridden
  No associated symptoms
  Moderate:Daily activities significantly restricted and most of the day patient is bedridden with or without associated symptoms
  Severe:Daily activities completely restricted, patient is bedridden all the day and always with associated symptoms
Lybecker score | 30 hours
  Mild
  Mild:Daily activities slightly restricted. Patient is not bedridden
  No associated symptoms
  Moderate:Daily activities significantly restricted and most of the day patient is bedridden with or without associated symptoms
  Severe:Daily activities completely restricted, patient is bedridden all the day and always with associated symptoms
Lybecker score | 36 hours
  Mild
  Mild:Daily activities slightly restricted. Patient is not bedridden
  No associated symptoms
  Moderate:Daily activities significantly restricted and most of the day patient is bedridden with or without associated symptoms
  Severe:Daily activities completely restricted, patient is bedridden all the day and always with associated symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A Hamed, MD, Principal Investigator — Faculty of medicine,Fayoum University
Locations (1):
- Fayoum University hospital, El Fayoum Qesm, Faiyum Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided